CLINICAL TRIAL: NCT03415607
Title: Comparison on Succinylcholine Onset Time Assessed by Train of Four Stimulation Versus Clinical Judgment During Rapid Sequence Induction
Brief Title: Comparison on Succinylcholine Onset Time Assessed by Train of Four Stimulation Versus Clinical Judgment During Rapid Sequence Induction of Anesthesia
Acronym: CELOTOF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: CELOTOF
Record Dates: First submitted 2018-01-16; First posted 2018-01-30 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2017-11

CONDITIONS: Suxamethonium Sensitivity; Aspiration of Gastric Contents Into Respiratory Tract, Part Unspecified
MeSH Terms: conditions — Butyrylcholinesterase deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Succinylcholine is a myorelaxant agent often used during rapid sequence induction for patients who need to undergo general anesthesia but who are at risk of pulmonary aspiration of gastric content. Whereas other myorelaxant agents are monitored with train of four stimulation to assess onset and duration, few anesthesiologists use train of four stimulation for onset of succinylcholine, as the anesthesiologists evaluate the effect with the time from injection (usually one minute) and the muscle fasciculation due to the release of acetylcholine.

The data available on onset duration of this drug are old and bases on only few studies, but the succinylcholine if sometime harmful (anaphylaxis , cardiac arrest, bronchospasm).

The investigators want to assess the onset time of succinylcholine with an objective toll , the train of four stimulation, and evaluate if the clinical judgment of the anesthesiologist is reliable to predict an adequate moment for endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Every patient undergoing general anesthesia with the use of suxamethonium for induction as assessed by the anesthesiologist

Exclusion Criteria:

* Patient under 18 years old
* Pregnant woman
* Nasotracheal intubation
* Monitoring of train of four at the adductor pollis impossible (such as patient with no arm )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patients undergoing general anesthesia with the use of suxamethonium for induction as assessed by the anesthesiologist
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Onset of action of suxamethonium as assessed by the measurement of the train of four stimulation at the adductor pollis | 60 seconds after the injection of suxamethonium
  Time, in seconds, between injection of suxamethonium and appearance of a value of zero on the train of four stimulation measurement (going to for on for to zero on for).
Time from suxamethonium injection to laryngoscopy | 60 seconds after the injection of suxamethonium
  Time, in seconds, between the injection of suxamethonium and the laryngoscopy realized by the anesthesiologist.

SECONDARY OUTCOMES:
Number of patients whom train of four was not 0 when they benefited from the laryngoscopy | 60 seconds after the injection of suxamethonium
Complications associated with use of suwamethnonium or early laryngoscopy | 60 seconds after the injection of suxamethonium
Main characteristics of the patients and intubation conditions | 60 seconds after the injection of suxamethonium

CONTACTS AND LOCATIONS:
Overall Officials: Clément Buléon, Principal Investigator — University Hospital, Caen
Locations (1):
- CHU Caen, Caen, France